CLINICAL TRIAL: NCT03786640
Title: Long Term Follow-up of the Tendril STS and Isoflex Leads in Conjunction With the Assurity MRI™ and Endurity MRI™ Pacemakers Within the 3T MRI Environment (Brady 3T MRI PMCF)
Brief Title: Abbott Brady 3T MRI PMCF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10266
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Syncope; Presyncope; Fatigue; Disorientation; Arrythmia; Bradycardia
Keywords: 3 Tesla MRI
MeSH Terms: conditions — Syncope; Fatigue; Confusion; Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Patients implanted with an SJM Tendril STS 2088 or Isoflex 1944/1948 lead, together with an Assurity MRI or Endurity MRI pacemaker, and who will undergo a 3T MRI scan are eligible to participate in this study.
  Interventions: Radiation: 3T MRI scan

INTERVENTIONS:
Radiation: 3T MRI scan — A clinically indicated 3T MRI scan will be performed per standard procedures for the radiology department. Cardiac monitoring during the MRI scan is recommended to include Pulse Oximetry and/or ECG.

SUMMARY:
The objective of this post-market, clinical follow up (PMCF) study, is to confirm the long-term safety of the Tendril STS and Isoflex leads, implanted with the Assurity MRI™ or Endurity MRI™ pacemakers, in patients undergoing a clinically indicated 3T MRI (3 Tesla Magnetic Resonance Imaging) scan.

DETAILED DESCRIPTION:
This prospective, non-randomized, observational study will be conducted at 35 centers worldwide where the study devices have 3T MR Conditional labeling; up to 110 patients will be enrolled, and will satisfy the recent PMCF requirement to maintain the CE mark.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be willing and able to provide informed consent for study participation (legal guardian or legally authorized representative is NOT acceptable).
2. Subject must be implanted with a St. Jude Medical Tendril STS 2088 or Isoflex 1944/1948 lead, and Assurity MRI or Endurity MRI pacemaker.
3. Capture threshold is stable and < 2.5V @ 0.5ms at the time of enrollment.
4. Subject is clinically indicated for a 3T MRI scan without sedation NOTE: Antianxiety agents (e.g. minor tranquilizers, etc.) may be used as long as the patient can communicate with site personnel during the MRI scan
5. Subject is willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

Exclusion Criteria:

1. The subject is currently participating in a clinical investigation that includes an active treatment arm that may confound the results of this study as determined by Abbott.
2. The subject is <18 years old (pediatric).
3. That subject has a life expectancy of less than 12 months due to any condition.
4. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
5. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
6. Any contraindication to MRI scan, including the presence of additional hardware (e.g. lead extenders, lead adapters, surgical staples, stents, dental braces, or abandoned leads).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with an SJM Tendril STS 2088 or Isoflex 1944/1948 lead, together with an Assurity MRI or Endurity MRI pacemaker, and who will undergo a 3T MRI scan are eligible to participate in this study. Subjects must meet all eligibility criteria and provide written informed consent prior to conducting any study procedures not considered standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a capture threshold increase of ≤ 0.5V at the permanently programmed pulse width | from pre- MRI scan to one-month post MRI scan

SECONDARY OUTCOMES:
Proportion of subjects with a sensing amplitude decrease of ≤ 50% from pre-MRI scan to one-month post-MRI scan | from pre-MRI scan to one-month post-MRI scan

OTHER OUTCOMES:
Rate of MRI-related adverse events | from pre- to 12-month post- MRI scan
  including but not limited to, the following:
  * Device (pulse generator) heating resulting in tissue damage in the implant pocket, or patient pocket discomfort, or both.
  * Induced currents on leads resulting in continuous capture, VT/VF, hemodynamic collapse, or all three.
  * Loss of pacing or capture in the MRI environment.

CONTACTS AND LOCATIONS:
Locations (9):
- Tartu University Hospital, Tartu, Estonia
- France (2):
  - Hopital Cardiovasculaire et Pneumologique Louis Pradel, Lyon, Auvergne-Rhône-Alpes
  - CHRU Hopital de Pontchaillou, Rennes, Brittany Region
- India (3):
  - Care Institute of Medical Sciences, Ahmedabad, Gurarat
  - Eternal Haert Care Centre, Jaipur, Rajasthan
  - Apollo Hospital, Chennai, Tamil Nadu
- AOU Federico II - Università degli Studi di Napoli, Napoli, Campania, Italy
- Netherlands (2):
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Albert Schweiter Ziekenhuis, Dordrecht, South Holland